CLINICAL TRIAL: NCT02105220
Title: Chest Wall Influence on Respiratory System Mechanics in Morbidly Obese Patients
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, PhD RRT, Massachusetts General Hospital
Other Study IDs: 2013P001413
Record Dates: First submitted 2014-02-12; First posted 2014-04-07 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Intra-Abdominal Hypertension
Keywords: Respiratory mechanics; Esophageal pressure; Functional residual capacity; positive end-expiratory pressure
MeSH Terms: conditions — Obesity; Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese: We will enroll patients with BMI≥40 kg/m2 to describe the impact of obesity on chest wall compliance and respiratory mechanics.
  Respiratory mechanics assessment: We will assess respiratory mechanics through different end expiratory pressure settings and recording airway and esophageal pressure tracings.
  Interventions: Other: Respiratory mechanics assessment
- Intraabdominal Hypertension: We will enroll patients with IAP≥12 mmHg to describe the impact of intraabdominal hypertension on chest wall compliance and respiratory mechanics.
  Respiratory mechanics assessment: We will assess respiratory mechanics through different end expiratory pressure settings and recording airway and esophageal pressure tracings.
  Interventions: Other: Respiratory mechanics assessment

INTERVENTIONS:
Other: Respiratory mechanics assessment — Data collection on respiratory mechanics, end expiratory lung volumes, gas exchanges, work of breathing. Data will be obtained by setting different end expiratory pressures and recording esophageal and airways pressure tracings.

SUMMARY:
The goal of this study is to describe the influence of the chest wall on the respiratory system mechanics in morbidly obese patients and in patients with high intra-abdominal pressure.

The effects of increasing and decreasing positive end-expiratory pressure (PEEP) on chest wall and total respiratory system mechanics, lung volumes and gas exchange will be evaluated, both during controlled and assisted mechanical ventilation.

Patients will be studied, first, during the acute phase of respiratory failure, when requiring intubation and controlled mechanical ventilation. Then, patients will be evaluated again during weaning from the ventilator to assess the influence of PEEP in assisted ventilation prior to extubation.

DETAILED DESCRIPTION:
The goal of this study is to describe the influence of the chest wall on the respiratory system mechanics. Investigators want to describe how extreme obesity and Intra-Abdominal Hypertension (IAH) affect normal respiratory system behavior. The effects of increasing and decreasing positive end-expiratory pressure (PEEP) on respiratory system mechanics, lung volumes and gas exchange will be evaluated, both during controlled and assisted mechanical ventilation.

Investigators will record and compare lung volumes, airway and transpulmonary pressure, gas exchange and hemodynamic changes caused by variations of PEEP. Patients will be studied, first, during the acute phase of respiratory failure, when requiring intubation and controlled mechanical ventilation. Patients will then again be evaluated during weaning from the ventilator to assess the influence of PEEP in assisted ventilation prior to extubation.

Investigators believe that assessment of the transpulmonary pressure and lung volumes is essential to correctly evaluate respiratory system function in patients in which the relationship between the lung and chest wall is altered. Improper mechanical ventilation leads to lung damage. High ventilatory volume/pressure are associated with lung overdistension, while low volume/pressure leads to lung collapse and cyclic opening and closing of alveoli. All of these mechanisms have been associated with ventilator induced lung injury and poorer outcomes. Adequate PEEP and transpulmonary pressure are fundamental in preventing this vicious cycle.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Requiring intubation and mechanical ventilation
* BMI≥40 kg/m2 or IAP≥12 mmHg

Exclusion Criteria:

* Known presence esophageal varices
* Recent esophageal trauma or surgery
* Severe thrombocytopenia (PTL≤10,000/mm3)
* Severe coagulopathy (INR≥2)
* Presence of pneumothorax
* Pregnancy
* Patients with diagnosed moderate to severe ARDS or with poor oxygenation index (PaO2/FiO2 < 200 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll morbidly obese intubated patients and/or patients affected by intraabdominal hypertension admitted to medical ICUs and surgical ICUs at Massachusetts General Hospital. Patients with contraindication to esophageal balloon placement or with severe respiratory failure will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
End Expiratory Lung Volumes | 2 hours
  EELV variation at different levels of PEEP in mechanically ventilated and sedated morbidly obese patients and patients with intraabdominal hypertension

SECONDARY OUTCOMES:
Respiratory mechanics | 24 hours
  Evaluation of effects of PEEP level set by ICU staff on respiratory mechanics after 24 hours from enrollment Evaluation of PEEP level set by ICU staff
Work of breathing | 20 minutes
  Evaluation of work of breathing variation at different level of PEEP during spontaneous breathing and ventilation weaning in morbidly obese patients
Respiratory mechanics | 2 hours
  Respiratory mechanics variation at different levels of PEEP in mechanically ventilated and sedated morbidly obese patients and patients with intraabdominal hypertension
Gas Exchange | 2 hours
  Gas exchange variation at different levels of PEEP in mechanically ventilated and sedated morbidly obese patients and patients with intraabdominal hypertension
Respiratory mechanics | 20 minutes
  Evaluation of respiratory mechanics at different level of PEEP during spontaneous breathing and ventilation weaning in morbidly obese patients
Gas exchange | 20 minutes
  Evaluation of gas exchange variation at different level of PEEP during spontaneous breathing and ventilation weaning in morbidly obese patients
End Expiratory Lung Volume | 24 hours
  Evaluation of effects of PEEP level set by ICU staff on EELV after 24 hours from enrollment
Gas Exchange | 24 hours
  Evaluation of effects of PEEP level set by ICU staff on gas exchange after 24 hours from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kacmarek, PhD RRT, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States